CLINICAL TRIAL: NCT02441140
Title: Detection of Tumor Associated Cell-free DNA in Peritoneal Fluid Obtained by Culdocentesis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Celula, Inc. (Industry)
Responsible Party: Principal Investigator, Neil S. Horowitz, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-029
Record Dates: First submitted 2015-04-14; First posted 2015-05-12 (Estimated); Last update posted 2020-05-04 (Actual); Status verified 2020-05

CONDITIONS: Stage III Ovarian Cancer; Stage IV Ovarian Cancer
Keywords: Stage III Ovarian Cancer; Stage IV Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paracentesis; Blood Specimen Collection; Tissue Banks

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Culdocentesis (Experimental): * Patients with known or highly likely ovarian cancer (i.e. highly elevated CA-125, ascites, pelvic mass) scheduled for cytoreductive surgery will be identified during preoperative consultation and offered participation in the study.
  * During Surgery:
    * Blood Collection
    * Vaginal Swab
    * Chromopertubation
    * Culdocentesis
    * Tissue Collection
  Interventions: Procedure: Culdocentesis; Procedure: Vaginal Swab; Procedure: Chromopertubation; Procedure: Blood collection; Procedure: Tissue collection

INTERVENTIONS:
Procedure: Culdocentesis — A sterile speculum will be placed in the vagina and the cervix identified. The cervix will be elevated using a tenaculum and a spinal needle inserted through the posterior vaginal fornix. Fluid from the posterior cul de sac will be collected
Procedure: Vaginal Swab — . A sterile speculum will be placed in the vagina and a Pap smear spatula will be used to swab the posterior fornix of the vagina. This swab will then be rinsed in a tube of saline.
Procedure: Chromopertubation — Chromopertubation is a common gynecologic technique used to test the patency of fallopian tubes during infertility evaluations. Fluid is flushed through the cervix and uterus and out the fallopian tubes.
Procedure: Blood collection — Intravenous blood collection will be drawn from an IV
Procedure: Tissue collection — As part of the standard surgical procedure for presumed ovarian cancer, the primary tumor will be resected and a sample obtained for evaluation

SUMMARY:
This research study is studying a possible test which may help doctors diagnose women with ovarian cancer.

DETAILED DESCRIPTION:
This research study is a Feasibility Study, to try to evaluate whether or not culdocentesis can detect tumor associated cell free DNA. Although this is the first time investigators are using this type of procedure to detect cell free DNA, culdocentesis is not a new procedure. It used to be done routinely in the past to examine pelvic fluid. The investigator's goal is to develop a test to detect ovarian cancer in women before they develop any signs or symptoms of the disease. Currently, there is no screening test for ovarian cancer.

This study uses a technique called "culdocentesis" to detect DNA released by ovarian cancer cells into pelvic fluid. During culdocentesis, a small needle is inserted through the vagina into an empty space between the uterus and the rectum called the "cul-de-sac." Fluid is withdrawn from this space and sent for analysis. Culdocentesis is a technique that has been used for many years to examine pelvic fluid and determine its composition, but it has not previously been studied as a technique for examining cell-free DNA to detect ovarian cancer. The investigators suspect that this may be a useful way to detect cell-free DNA from ovarian cancer cells because the ovaries are very close to the cul-de-sac space.

In this study, the investigators will compare our ability to detect cell-free DNA in fluid from the cul-de-sac with our ability to detect cell-free DNA from a vaginal swab (similar to a Pap smear), a blood test, and in the tissue specimens collected at the time of surgery. The investigators are hoping to learn from this study whether developing a cell-free DNA test to screen for ovarian cancer involving culdocentesis would be an effective strategy.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age ≥ 18
* Able to give informed consent
* Scheduled for surgery at Brigham and Women's Hospital for known or highly suspected Stage III or IV ovarian cancer (i.e. elevated CA-125 with a pelvic mass, ascites, and carcinomatosis)
* Post-menopausal or negative urine and/or blood pregnancy test
* Measurable disease on preoperative imaging

Exclusion Criteria:

* Male
* Age < 18
* Unable to give informed consent
* Not planned for surgical intervention
* Active malignancy other than ovarian cancer
* Prior bilateral tubal ligation or hysterectomy (as this would prevent chromopertubation)
* Known or suspected active pelvic infection
* Pregnancy
* No measurable disease or suspected Stage I or II ovarian cancer on preoperative imaging

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-05; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Number of completed peritoneal fluid collection by culdocentesis after chromopertubation as an assessment of feasibility of peritoneal fluid collection in women with ovarian cancer. | At the time of surgery

SECONDARY OUTCOMES:
Measure the concentration of cell free DNA in various biologic fluids and compare it to primary tumor DNA. | At the time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Neil Horowitz, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts